CLINICAL TRIAL: NCT01068782
Title: A Phase 2 Non-Comparative Randomized Open-Label Study of Multiple Regimens of Single-Agent XL184 in Subjects With Grade IV Astrocytic Tumors in First or Second Relapse
Brief Title: Study of Multiple Doses and Regimens of XL184 (Cabozantinib) in Subjects With Grade IV Astrocytic Tumors in First or Second Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL184-205
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Astrocytic Tumors
Keywords: Glioblastoma; Glioma; Brain Cancer; Brain Tumor; Astrocytoma
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms; Astrocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: XL184
- Arm 2 (Experimental)
  Interventions: Drug: XL184
- Arm 3 (Experimental)
  Interventions: Drug: XL184
- Arm 4 (Experimental)
  Interventions: Drug: XL184

INTERVENTIONS:
Drug: XL184 — given orally as capsules

SUMMARY:
This is a study of multiple regimens of single-agent XL184 in subjects with grade IV astrocytic tumor in first or second relapse. The Randomized Phase of the study will evaluate the safety, tolerability, and preliminary efficacy of four XL184 dosing regimens in separate study arms. Subjects will be randomized to one of the study arms, which will not be blinded. After the Randomized Phase, additional subjects will be enrolled to further expand one study arm in the Expansion Phase.

ELIGIBILITY:
Inclusion Criteria:

* The subject has histologically confirmed diagnosis at any time of grade IV astrocytic tumor as determined by the investigator. Tumor samples will be required for pathology review.
* The subject has received prior standard radiation for any grade astrocytic tumor.
* The subject has received prior temozolomide (Temodar) therapy
* The subject has had one or two progressions as grade IV astrocytic tumor from any grade, as determined by investigator
* The subject must have a qualifying brain MRI scan within a specific timeframe prior to start of study treatment
* For subjects with recent tumor resection or biopsy, starting on study must occur a specified amount of time after the surgery and the subject must have recovered from the effects of surgery
* The subject has a Karnofsky Performance Status ≥ 70% and has the ability to swallow whole capsules
* The subject is capable of understanding the informed consent and has signed the informed consent document
* The subject has adequate organ and marrow function
* Sexually active subjects (male and female) must agree to use medically accepted methods of contraception during the course of the study and for 6 months following discontinuation of study treatment
* The subject has had no other diagnosis of malignancy (certain exceptions apply)
* Female subjects of childbearing potential must have a negative pregnancy test at screening

Exclusion Criteria:

* The subject has received certain prior anticancer therapies within a certain amount of time before starting study treatment
* The subject is receiving warfarin (or other coumarin derivatives) and is unable to switch to low molecular weight heparin
* The subject has evidence of acute intracranial or intratumoral hemorrhage either by MRI or CT scan. Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin are eligible
* The subject is unable to undergo MRI scan (eg, has pacemaker)
* The subject has received enzyme-inducing anti-epileptic agents within a certain time prior to starting study treatment (eg, carbamazepine, phenytoin, phenobarbital, primidone)
* The subject has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 Grade ≤ 1 from AEs (except alopecia and lymphopenia) due to surgery, or other medications that were administered prior to study start
* The subject has evidence of unhealed wounds
* The subject is pregnant or breast-feeding
* The subject has serious intercurrent illness or a recent history of serious disease
* The subject has inherited bleeding diathesis or coagulopathy (disease affecting how blood clots) with the risk of bleeding
* The subject has a history of any medical or surgical conditions (eg, stomach or intestinal surgery or resection) that would potentially interfere with or alter gastrointestinal function
* The subject has a history of idiopathic pulmonary fibrosis or interstitial lung disease
* The subject has received any live virus vaccine or any inactivated vaccine within a certain amount of time before starting study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
In the Randomized Phase, to evaluate the preliminary efficacy and tolerability of multiple regimens of XL184 | Assessed every 1-3 weeks, during study visits
In the Expansion Phase, to evaluate the efficacy of XL184 treatment | Assessed every 6 weeks

SECONDARY OUTCOMES:
To further evaluate the safety and tolerability of XL184 treatment during the entire treatment period | Assessed every 1-3 weeks, during study visits
To further characterize the pharmacokinetic and pharmacodynamic parameters of XL184 | Assessed every 3-4 weeks, during study visits

CONTACTS AND LOCATIONS:
Locations (17):
- United States (15):
  - Birmingham, Alabama
  - Encinitas, California
  - Pleasant Hill, California
  - Chicago, Illinois
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Amhearst, New York
  - Rochester, New York
  - Cleveland, Ohio
  - Hershey, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Seattle, Washington
- Canada (2):
  - Calgary, Alberta
  - Montreal, Quebec